CLINICAL TRIAL: NCT00363207
Title: Behavior of Children in the Following Appointment Related to Numbness Perception After Dental Local Anesthesia
Brief Title: Behavior of Children Related to Numbness After Dental Local Anesthesia
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Diana Ram, Hadassah Medical Organization
Other Study IDs: STDI-HMO-CTIL
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2007-04

CONDITIONS: Anesthesia, Local; Anesthesia, Dental
Keywords: behavior; local anesthesia; behavior after dental local anesthesia
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In children, behavior management is critical to the success of pediatric dental procedures. Most of the studies on local anesthesia performed in children deal with the question how to avoid or minimize pain during injection. Due to the sensation of numbness children scratch the soft tissues and bite lips and tongue. In many cases, this may be kept in children's memory as a "painful experience" and may affect their behavior in the following visit. The purpose of this study is to evaluate children's reactions to the administration of local anesthetic injection in the mandible (mandibular block) and in the maxilla (supraperiosteal infiltration), and to assess their behavior in the following visit related to each type of injection.

DETAILED DESCRIPTION:
Children between the ages of 4 to 7, undergoing dental treatment at the Department of Pediatric dentistry of the Hadassah School of Dental Medicine will participate in the study. All patients should be ASA Class I with no prior dental treatment who need at least two clinical sessions of similar operative procedures preceded by local anesthetic injection, one in each jaw, none of which due to emergency. Subjective and objective evaluation will be performed according to previously validated scales.

ELIGIBILITY:
Inclusion Criteria:

* Age: 4-7
* Behavior: Frankel 3-4
* No sedation (premedication)
* ASA 1
* No dental treatment before
* Need for similar treatment in the upper and lower jaw
* No emergency treatment

Exclusion Criteria:

* Need of premedication
* Uneven treatment in each jaw

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children receiving routine dental treatment at the hadassah school of dental medicine
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-05; Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Ram, Dr, Principal Investigator — Hadassah Medical Organization
Locations (2):
- Israel (2):
  - Hadassah School of Dental Medicine, Jerusalem, Jerusalem
  - Hadassah Medical Organization, Jerusalem